CLINICAL TRIAL: NCT00836017
Title: CD-PROBE: Cervical Dystonia Patient Registry for the Observation of onabotulinumtoxinA Efficacy
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MedAff BTX-0718
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-06

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BOTOX®: Patients received BOTOX® (onabotulinumtoxinA) treatment as standard of care in clinical practice as prescribed by the physician. No intervention was administered as part of the study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention was administered as part of the study.

SUMMARY:
This study is an observational trial which will measure the efficacy of onabotulinumtoxinA in treating Cervical Dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cervical Dystonia
* Candidate for botulinum toxin type A therapy
* New to physician's practice, and/or new to botulinum toxin type A therapy, or has not been injected with botulinum toxin type A for at least 16 weeks as a participant in another clinical trial investigating botulinum toxin type A for cervical dystonia
* Able to follow study instructions and complete study activities

Exclusion Criteria:

* Patients undergoing elective surgery during the trial period
* Females who are pregnant, nursing, or planning a pregnancy
* History of poor cooperation or compliance with medical treatment or unreliability
* Any condition or situation in which, in the investigator's opinion, places the patient at significant risk, could confound the study data, or may interfere with the patient's participation in the study, including but not limited to unstable medical conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cervical Dystonia whom are being treated with onabotulinumtoxinA
Sampling Method: Non-Probability Sample
Enrollment: 1046 (Actual)
Dates: Start 2009-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Springfield, Massachusetts, United States

REFERENCES:
- [Derived] Agarwal P, Barbano R, Moore H, Schwartz M, Zuzek A, Sadeghi M, Patel A. OnabotulinumtoxinA Dosing, Disease Severity, and Treatment Benefit in Patients With Cervical Dystonia: A Cohort Analysis From CD PROBE. Front Neurol. 2022 Jun 30;13:914486. doi: 10.3389/fneur.2022.914486. eCollection 2022. PMID 35847221
- [Derived] Molho ES, Stacy M, Gillard P, Charles D, Adler CH, Jankovic J, Schwartz M, Brin MF. Impact of Cervical Dystonia on Work Productivity: An Analysis From a Patient Registry. Mov Disord Clin Pract. 2016 Mar-Apr;3(2):130-138. doi: 10.1002/mdc3.12238. Epub 2015 Dec 16. PMID 27774495
- [Derived] Jankovic J, Adler CH, Charles D, Comella C, Stacy M, Schwartz M, Manack Adams A, Brin MF. Primary results from the cervical dystonia patient registry for observation of onabotulinumtoxina efficacy (CD PROBE). J Neurol Sci. 2015 Feb 15;349(1-2):84-93. doi: 10.1016/j.jns.2014.12.030. Epub 2014 Dec 27. PMID 25595221
- [Derived] Jankovic J, Adler CH, Charles PD, Comella C, Stacy M, Schwartz M, Sutch SM, Brin MF, Papapetropoulos S. Rationale and design of a prospective study: Cervical Dystonia Patient Registry for Observation of OnaBotulinumtoxinA Efficacy (CD PROBE). BMC Neurol. 2011 Nov 4;11:140. doi: 10.1186/1471-2377-11-140. PMID 22054223

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BOTOX®
Started | 1046
Completed | 502
Not Completed | 544

BASELINE CHARACTERISTICS:
Population: Baseline measures were based on all enrolled participants who received treatment.
Arm/Group | BOTOX®
Number analyzed (Participants) | 1041
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 774
  Male | 267

OUTCOME MEASURES:

1. Primary Outcome: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Total Score
Description: TWSTRS is an assessment scale used to measure the impact of cervical dystonia on patients. The score is comprised of 3 subscales: Severity, Disability, and Pain, each of which is scored independently. The total of these 3 subscales comprises the TWSTRS total score which is scored from 0 (least symptoms) to 85 (worst symptoms). Higher scores indicate a greater degree of symptom severity.
Time Frame: 4-6 weeks after treatment 3 (Up to 104.3 weeks)
Population: All participants with data available for this outcome measure at all visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BOTOX®
Number analyzed (Participants) | 479
score on a scale | 27.1 (14.6)

2. Secondary Outcome: Percentage of Participants With Cervical Dystonia (CD) Severity Mild
Description: The physician assessed the patient's severity of CD using a 3-point scale: mild, moderate or severe. The percentage of participants with CD Severity Mild is reported.
Time Frame: Baseline, 4-6 weeks after treatment 3 (Up to 104.3 weeks)
Population: All participants with data available for this outcome measure at all visits.
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX®
Number analyzed (Participants) | 475
percentage of participants
  Baseline | 30.5
  4-6 weeks after treatment 3 | 58.5

3. Secondary Outcome: Percentage of Participants With Improvement in Clinicians Global Impression of Change
Description: The physician evaluated the change in the patient's present condition compared to Baseline using a 7-point scale where: 1= very much improved to 7= very much worse. The percentage of participants where the physician's response was: 1=very much improved, 2=much improved or 3=minimally improved is reported.
Time Frame: Baseline, 4-6 weeks after treatment 3 (Up to 104.3 weeks)
Population: All participants with data available for this outcome measure at all visits.
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX®
Number analyzed (Participants) | 479
percentage of participants | 95.0

4. Secondary Outcome: Percentage of Participants With Improvement in the Patient Global Impression of Change
Description: The patient evaluated the change in their present condition compared to Baseline using a 7-point scale where: 1= very much improved to 7= very much worse. The percentage of participants with responses: 1=very much improved, 2=much improved or 3=minimally improved is reported.
Time Frame: Baseline, 4-6 weeks after treatment 3 (Up to 104.3 weeks)
Population: Participants with data available for this outcome measure at all visits.
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX®
Number analyzed (Participants) | 470
percentage of participants | 91.7

5. Secondary Outcome: Pain Numeric Rating Scale Score
Description: Patients rated their level of pain during the past 24 hours using an 11-point scale where: 0=no pain to 10= pain as bad as you can imagine. A lower number score indicated a lower amount of pain.
Time Frame: Baseline, 4-6 weeks after treatment 3 (Up to 104.3 weeks)
Population: Participants with data available for this outcome measure at all visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BOTOX®
Number analyzed (Participants) | 286
score on a scale
  Baseline | 6.2 (2.2)
  4-6 weeks after treatment 3 | 4.2 (2.5)

ADVERSE EVENTS:
Description: The number of participants at risk for Serious Adverse Events and Adverse Events was based on all enrolled participants who received treatment.
Arm/Group | BOTOX®
Serious Adverse Events (participants affected / at risk) | 33/1041
Other Adverse Events (participants affected / at risk) | 138/1041
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=1041)
Cardiac arrest (Cardiac disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Intestinal mass (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Pyrexia (General disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 2
Overdose (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Mental disorder (Psychiatric disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Alcohol detoxification (Surgical and medical procedures) | 1
Cardiac operation (Surgical and medical procedures) | 1
Tracheostomy tube removal (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=1041)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 73
Dysphagia (Gastrointestinal disorders) | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.